CLINICAL TRIAL: NCT03683511
Title: Population Pharmacokinetics Modeling : a Priori Optimization of Amikacin First Dose in Critically Ill Patients Using a Nomogram
Brief Title: Nomograms for Optimization of Amikacin First Dose in Critically Ill Patients Using a Population Pharmacokinetics Model
Acronym: PIC-AMI
Status: Completed | Type: Observational
Sponsor: Nantes University Hospital (Other)
Collaborators: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: RC14_0121
Record Dates: First submitted 2018-09-13; First posted 2018-09-25 (Actual); Last update posted 2018-09-25 (Actual); Status verified 2018-09

CONDITIONS: Pharmacokinetics
Keywords: amikacin

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to elaborate nomograms to optimize amikacine first dosing in critically ill patients, using a population pharmacokinetics model elaborated with multicentric data.

DETAILED DESCRIPTION:
French guidelines recommend for probabilistic therapy to reach an amikacin concentration 1 hour after beginning the infusion ≥ 60 mg/L. This target is rarely achieved in the ICU despite a 30 mg/kg recommended dosage. Using data collected prospectively in critically ill patients of Nîmes (France) (1) and Nantes (France), we will elaborate a population pharmacokinetic model on the non-parametric software Pmetrics and on the parametric software Monolix. We will calculate probability of target attainment of Monte-Carlo simulations, using the non-parametric model. Nomograms to determine optimal first dose of amikacin in critically ill patients, according to a few variables previously identified, will be produced.

ELIGIBILITY:
Inclusion Criteria:

* patients treated with amikacin for sepsis in one of the participating ICU will be included.

Exclusion Criteria:

* patients with aminoglycoside allergy, history of myasthenia, pregnancy, under guardianship.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated with amikacin for sepsis ou septic shock in the medical intensive care unit of Nantes,France or in an ICU of Nîmes, France will be recruited.
Sampling Method: Non-Probability Sample
Enrollment: 138 (Actual)
Dates: Start 2014-04-21 (Actual); Primary Completion 2016-06-30 (Actual); Study Completion 2016-06-30 (Actual)

PRIMARY OUTCOMES:
amikacin infusion | one hour after beginning of infusion.ed
  Target is defined as 8 times x Minimal Inhibatory Concentration for MIC = 4 mg/L and MIC = 8 mg/L. Those PTA will be calculated using the final pharmacokinetics model, according to the dependent variables.

SECONDARY OUTCOMES:
maximal dose of amikacin (in mg) allowed to have a probability of target attainment (PTA) of 50% or less for the trough concentration. | 24 hours after beginning of infusion
  Target is 2.5 mg/L. Those PTA will be calculated using the final pharmacokinetics model, according to the dependent variables.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Nantes, Nantes, France

REFERENCES:
- [Background] Roger C, Nucci B, Louart B, Friggeri A, Knani H, Evrard A, Lavigne JP, Allaouchiche B, Lefrant JY, Roberts JA, Muller L. Impact of 30 mg/kg amikacin and 8 mg/kg gentamicin on serum concentrations in critically ill patients with severe sepsis. J Antimicrob Chemother. 2016 Jan;71(1):208-12. doi: 10.1093/jac/dkv291. Epub 2015 Oct 1. PMID 26429564